CLINICAL TRIAL: NCT05714605
Title: Implementation and Evaluation of THRIVE: A Health Innovation to Support Care Transitions for Medicaid-Insured Individuals Following Hospitalization
Brief Title: Implementation and Evaluation of A Health Innovation to Support Medicaid-Insured Individuals Following Hospitalization
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Rita & Alex Hillman Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10080229
Record Dates: First submitted 2023-01-19; First posted 2023-02-06 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Care Transitions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THRIVE Intervention (Experimental): 1 month intensive post discharge case management and care coordination.
  Interventions: Behavioral: THRIVE Intervention
- Usual Care (No Intervention): Discharge to home without intensive post acute case management or care coordination.

INTERVENTIONS:
Behavioral: THRIVE Intervention — The THRIVE Clinical Pathway is a standardized transitional care clinical pathway that supports Medicaid insured or Medicaid eligible individuals following hospitalization.
  Arms: THRIVE Intervention

SUMMARY:
The goal of this stepped wedge pragmatic trial is to compare referral patterns and post discharge outcomes in Medicaid insured individuals discharge following a hospitalization]. The aims are to 1) evaluate the implementation of the THRIVE clinical pathway, including feasibility, appropriateness, and acceptability and 2) examine referral patterns, 30- day readmission and Emergency Department (ED) utilization patterns for participants who receive THRIVE support services. During hospitalization participants will receive a referral to home care services and will be seen by a home care nurse within 48 hours following discharge. A discharging physician or Advanced Practice Provider will maintain clinical oversight for 30 days or until the patient sees primary care provider or specialist. A Care Coordination Team conducts weekly case conferences to ensure social and health needs are being addressed for 30 days post-discharge. Researchers will compare Medicaid insured patients discharged during the study, to those receiving usual care to determine if there are differences in post-acute utilization outcomes.

DETAILED DESCRIPTION:
This is a prospective single site Type 1 hybrid effectiveness-implementation parallel mixed methods (QUANT + qual) quasi-experimental study. This study design involves simultaneous collection and analysis of quantitative and qualitative data, giving priority weight to the quantitative data to evaluate program referrals, outcomes, and program fidelity, while qualitative data will evaluate process through detailed descriptions of perspectives of barriers and facilitators faced by health care providers in implementing the THRIVE intervention. Qualitative interviews will also assess stakeholder perspectives of the value of the intervention in addressing health inequities among Medicaid insured individuals cared for in the acute and home care settings. Nesting the qualitative interview within a single-site randomized trial of a the THRIVE intervention will allow us to determine whether the intervention improved primary outcomes (referrals to homecare, 30-day readmission, ED utilization, connection to PCP) and to identify professional and organizational barriers to implementation. Combining these insights with that of effectiveness outcome date will allow consideration for meaningful contextual factors that are viewed as critical to the implementation of THRIVE and subsequent outcomes. Our stepped wedge design with include a randomized roll-out to case managers at Pennsylvania Hospital and the study will be carried out over 18 months. To begin, 5 case managers will be randomized to receive training on the THRIVE clinical pathway. Following training they will be invited to begin offering referrals to the THRIVE clinical pathway. After 2 months the remaining 4 case managers will be trained on the THRIVE intervention and will be able to begin submitting referrals.

ELIGIBILITY:
Inclusion Criteria:

* Medicaid insured
* Residing in the state of Pennsylvania
* Experienced a hospitalization at study hospital
* Agrees to home care at partner home care setting.

Exclusion Criteria:

* Individuals under age 18

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rates of Referrals to Homecare | Through study completion, an average of 18 months
  We will evaluate changes in home care referrals between case managers exposed to the intervention compared to those who were not.
Rates of Readmissions | 30 days following hospital discharge
  We will evaluate the rate of readmissions over the course of the study for THRIVE participants compared to those receiving usual care.
Rates of Emergency Department Visit | 30 days following hospital discharge
  We will evaluate the rate of ED visits over the course of the study for THRIVE participants compared to those receiving usual care.
Primary Care or Specialist Visit | 30 Days following hospital discharge
  We will compare the rates of primary care provider and specialist visits within 30 days following discharge compared to those receiving usual care.

SECONDARY OUTCOMES:
Feasibility, Acceptability, Appropriateness, Workload | Through study completion, an average of 18 months
  We will conduct interviews of clinicians at the conclusion of the study to gather perceptions of the THRIVE clinical pathway and facilitators and barriers to engaging with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Margo B Brooks Carthon, PhD RN, Principal Investigator — University of Pennsylvania
Locations (1):
- Pennsylvania Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brooks Carthon JM, Brom H, Grantham-Murrillo M, Sliwinski K, Mason A, Roeser M, Miles D, Garcia D, Bennett J, Harhay MO, Flores E, Amenyedor K, Clark R. Equity-Centered Postdischarge Support for Medicaid-Insured People: Protocol for a Type 1 Hybrid Effectiveness-Implementation Stepped Wedge Cluster Randomized Controlled Trial. JMIR Res Protoc. 2024 Mar 26;13:e54211. doi: 10.2196/54211. PMID 38530349